CLINICAL TRIAL: NCT02764112
Title: Assessing the Ability of Warfarin Treated Patients to Predict Their INR
Status: Completed | Type: Observational
Sponsor: Northeast Iowa Medical Education Foundation (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Principal Investigator, Jim Hoehns, Research Director, Northeast Iowa Medical Education Foundation
Other Study IDs: 914
Record Dates: First submitted 2016-03-30; First posted 2016-05-06 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
Keywords: warfarin
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
ASSESSING THE ABILITY OF WARFARIN TREATED PATIENTS TO PREDICT THEIR INR Kathleen McNamara, James Hoehns, Matthew Witry

The international normalized ratio (INR) is the accepted lab test used to measure the intensity of warfarin effect. The conventional wisdom is that patients receiving warfarin are unable to correctly determine, in the absence of an INR result, whether or not they are therapeutic at any given time. Some warfarin treated patients express that they have insight into what their INR result will be. Various patient related factors may contribute to these opinions.

Our objective is to assess how accurately patients can guess their INR result before it is obtained and to describe factors which inform their opinion of what their INR will be.

DETAILED DESCRIPTION:
ASSESSING THE ABILITY OF WARFARIN TREATED PATIENTS TO PREDICT THEIR INR Kathleen McNamara, James Hoehns, Matthew Witry

The international normalized ratio (INR) is the accepted lab test used to measure the intensity of warfarin effect. The conventional wisdom is that patients receiving warfarin are unable to correctly determine, in the absence of an INR result, whether or not they are therapeutic at any given time. Some warfarin treated patients express that they have insight into what their INR result will be. Various patient related factors may contribute to these opinions.

Our objective is to assess how accurately patients can guess their INR result before it is obtained and to describe factors which inform their opinion of what their INR will be. In this prospective study, the investigators will enroll warfarin treated patients from 7 anticoagulation clinics in Iowa. Inclusion criteria are: age ≥18 years, warfarin use ≥60 days, INR goal of 2.0-3.0 or 2.5-3.5, expected warfarin use >6 months, and English speaking. Exclusion criteria include: use of self INR-testing, home INR draws, dementia, or residing in a long-term care facility. A data collection form will be completed prior to INR measurement for a 6 month period. Information will be collected for subject demographics, warfarin adherence, INR stability, INR prediction, and prediction rationale.

INR monitoring represents a significant burden with respect to cost and time. The results of this study may identify patient factors which could help individualize and decrease the frequency of INR monitoring in patients who receive maintenance warfarin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Warfarin use ≥60 days
* INR goal of 2.0-3.0 or 2.5-3.5
* Expected warfarin use >6 months
* English speaking

Exclusion Criteria:

* Self INR-testing
* Home INR draws
* Dementia
* Residence of a long-term care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective study, we will enroll warfarin treated patients from 8 anticoagulation clinics in Iowa. Inclusion criteria are: age ≥18 years, warfarin use ≥60 days, INR goal of 2.0-3.0 or 2.5-3.5, expected warfarin use >6 months, and English speaking. Exclusion criteria include: use of self INR-testing, home INR draws, dementia, or residing in a long-term care facility.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Assess factors which influence INR predictions | 6 months
  Patients will be asked to predict their INR value prior to having it tested. We will record patient's INR prediction and the value we obtain after testing INR.

CONTACTS AND LOCATIONS:
Locations (1):
- Northeast Iowa Family Practice, Waterloo, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McNamara K, Witry M, Bryant G, Koenigsfeld C, Lehman N, Logemann C, Mormann M, Rueber A, Herring M, Hoehns JD. A prospective, multi-center cohort study: investigating the ability of warfarin-treated patients to predict their INR. Clin Res Cardiol. 2019 Feb;108(2):212-217. doi: 10.1007/s00392-018-1345-9. Epub 2018 Aug 8. PMID 30091085